CLINICAL TRIAL: NCT00838279
Title: Randomized, 2-Way Crossover, Bioequivalence Study of Lamotrigine 25 mg Chewable Dispersible Tablets and Lamictal® 25 mg Chewable Dispersible Tablets in Healthy Subjects Under Fasting Conditions
Brief Title: Lamotrigine 25 mg Chewable Tablets, Fasting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 01303
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lamotrigine (Experimental): Lamotrigine 2 x 25 mg Chewable Tablet (test) dosed in first period followed by Lamictal® 2 x 25 mg Chewable Tablet (reference) dosed in second period
  Interventions: Drug: Lamotrigine 25 mg Chewable Tablets
- Lamictal® (Active Comparator): Lamictal® 2 x 25 mg Chewable Tablet (reference) dosed in first period followed by Lamotrigine 2 x 25 mg Chewable Tablet (test) dosed in second period
  Interventions: Drug: Lamictal® 25 mg Chewable Tablets

INTERVENTIONS:
Drug: Lamotrigine 25 mg Chewable Tablets — 2 x 25 mg, single-dose fasting
  Arms: Lamotrigine
Drug: Lamictal® 25 mg Chewable Tablets — 2 x 25 mg, single-dose fasting
  Arms: Lamictal®

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of lamotrigine 25 mg chewable dispersible tablets (test) versus Lamictal® (reference) administered as 2 x 25 mg chewable dispersible tablets under fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be females and/or males, non-smokers, 18 years of age and older.
* Female subjects will be post-menopausal or surgically sterilized.
* Post-menopausal status is defined as absence of menses for the past 12 months or hysterectomy with bilateral oophorectomy at least 6 months ago.
* Sterile status is defined as hysterectomy, bilateral oophorectomy or tubal ligation at least 6 months ago.

Exclusion Criteria:

* Clinically significant illnesses within 4 weeks of the administration of the study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Subjects with a history of renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma, diabetes, psychosis or glaucoma will not be eligible for this study.
* Any reason which, in the opinion of the medical sub-investigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive urine drug screen at screening.
* Positive testing for hepatitis B, hepatitis C or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, or diastolic blood pressure lower than 50 or over 90; or heart rate less than 50 bpm) at screening.
* Subjects with BMI ≥ 30.0.
* History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than two units of alcohol per day (1 Unit - 150 mL of wine or 360 mL of beer or 45 mL of alcohol 40%).
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PVP) and crack) within 1 year of the screening visit.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the medical sub-investigator, contraindicates the subject's participation in this study.
* History of allergic reactions to lamotrigine.
* Use of any drugs known to induce or inhibit drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin; examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin, ketoconazole, MAO inhibitors, neuroleptics, verapamil, quinidine, valproic acid), use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural products, vitamins, garlic as supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Subjects who have had a depot injection or an implant of any drug 3 months prior to administration of study medication.
* Subjects who have dentures or braces.
* Donation of plasma (500 mL) within 7 days. Donation or loss of whole blood prior to administration of the study medication as follow: less than 300 mL of whole blood within 30 days; 300 mL to 500 mL of whole blood within 45 days; more than 500 mL of whole blood within 56 days.
* Positive alcohol breath test at screening.
* Subjects who have used tobacco in any form within 90 days preceding study drug administration.
* Female subjects: breast-feeding subjects.
* Female subjects: positive urine pregnancy test at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2002-02; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bicrell, M.D., Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc., Sainte-Foy, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Lamotrigine (Test) First: Lamotrigine 2 x 25 mg Chewable Tablet (test) dosed in first period followed by Lamictal® 2 x 25 mg Chewable Tablet (reference) dosed in second period
- Lamictal® (Reference) First: Lamictal® 2 x 25 mg Chewable Tablet (reference) dosed in first period followed by Lamotrigine 2 x 25 mg Chewable Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Lamotrigine (Test) First | Lamictal® (Reference) First
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Washout
Arm/Group | Lamotrigine (Test) First | Lamictal® (Reference) First
Started | 16 | 16
Completed | 15 | 15
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention
Arm/Group | Lamotrigine (Test) First | Lamictal® (Reference) First
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lamotrigine (Test) First | Lamictal® (Reference) First | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 15 | 16 | 31
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 13 | 12 | 25
  Black | 3 | 2 | 5
  American Hispanic | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence basd on Cmax
Time Frame: Blood samples collected over 120 hour period
Population: Two subjects did not complete the study, and there was an issue with dosing of one subject (the whole tablet was not consumed for one of the periods) therefore there are 29 data sets that were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Lamotrigine: Lamotrigine 2 x 25 mg Chewable Tablet (test) dosed in either period
- Lamictal®: Lamictal® 2 x 25 mg Chewable Tablet (reference) dosed in either period
Arm/Group | Lamotrigine | Lamictal®
Number analyzed (Participants) | 29 | 29
ng/mL | 713.46 (95.02) | 709.97 (84.37)
Statistical Analysis 1: Comparison: Lamotrigine vs Lamictal®; Test type: Non-Inferiority or Equivalence — Using GLM procedures in SAS, analysis of variance (ANOVA)was performed on log-transformed AUC0-t, AUC0-inf and Cmax at the significance level of 0.05; Test/Ref Ratio of LS Means x 100 = 100.31, 90% CI [97.82 to 102.85] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 120 hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Lamotrigine | Lamictal®
Number analyzed (Participants) | 29 | 29
ng*h/mL | 34541.03 (14354.41) | 33498.85 (12316.96)
Statistical Analysis 1: Comparison: Lamotrigine vs Lamictal®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 101.78, 90% CI [99.09 to 104.55] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 120 hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lamotrigine | Lamictal®
Number analyzed (Participants) | 29 | 29
ng/mL | 28843.06 (6866.12) | 28923.66 (7355.31)
Statistical Analysis 1: Comparison: Lamotrigine vs Lamictal®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 99.94, 90% CI [97.40 to 102.55] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.